CLINICAL TRIAL: NCT02256501
Title: Intracoronary Transplantation of Autologous Bone Marrow Derived Mononuclear Cells (MNC) in Idiopathic Dilated Cardiomyopathy in Pediatric Patients: Clinical Trial Phase I/II
Brief Title: Intracoronary Transplantation of Bone Marrow Derived Mononuclear Cells in Pediatric Cardiomyopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nasser Aghdami MD., PhD (Other Government)
Responsible Party: Sponsor-Investigator, Nasser Aghdami MD., PhD, Hear of department of Regenerative Medicine of Royan Institute 7 cell therapy center, Royan Institute
Organization: Royan Institute (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Heart-004
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Cardiomyopathy
Keywords: Dilated cardiomyopathy pediatric heart failure cell therapy
MeSH Terms: conditions — Cardiomyopathies | interventions — Transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mono Nunlear Cell (MNC) (Experimental): The patients with idiopathic dilated cardiomyopathy who underwent intracoronary injection of autologous bone marrow-derived mononuclear cells .
  Interventions: Biological: Mono Nuclear Cell (MNC) transplantation
- Control (No Intervention): The patients with cardiomyopathy that are under observe during the study.

INTERVENTIONS:
Biological: Mono Nuclear Cell (MNC) transplantation — Intracoronary administration of autologous bone marrow derived mononuclear cells
  Arms: Mono Nunlear Cell (MNC)

SUMMARY:
According to the high morbidity and mortality of idiopathic Dilated CardioMyopathy (IDCM) in pediatric, new modality of treatment is emerging. There are some case reports of administration of stem cell therapy. The investigators design the first randomized clinical trial in this setting. The investigators enroll 32 pediatric IDCM patients in two groups (16 pts. in each group including cell therapy and control). The investigators assess the safety and efficacy of intracoronary transplantation of autologous bone marrow derived mononuclear cells in this patients compared to control group.

DETAILED DESCRIPTION:
Dilated cardiomyopathy as the most common form of cardiomyopathy is a rare but life-threatening disorder in children. The primary cause of nearly 37 % of children with DCM was unknown at diagnosis. Despite of the developing in the medical and surgical treatment during the past several decades, standard treatments (including Digitalis, diuretics, inhibitors of ACE, beta blockers, antiplatelet drugs and treatments Antiarrhythmic), may stabilize the condition, but will not restore heart function to its previous condition. Therapy remains complex and expensive. For some not all children the heart transplantation is only option and mortality continues to be high, also. Stem cell and cell-based therapies offer an innovative approach to reverse cardiac structure and function towards normal, possibly reducing the need for aggressive therapies and cardiac transplantation. According to the inclusion and exclusion criteria of trial, 32 patients with left ventricular ejection fraction less than 45% who resistance to the standard medical therapy were randomly allocated in 2 groups including BM-derived mononuclear (n=16) and control (n=16). Only the MNC group underwent the bone marrow aspiration and intracoronary injection. The investigators followed all of patients at 2 weeks, 1, 2, 4 and 6 months after transplantation for cell therapy group or registration for placebo by physical examination, laboratory tests and imaging such as echocardiography, CXR and CMR.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1-16 year(s)
2. LVEF <45% (echocardiography)
3. Duration of diagnosis more than 3 months
4. Resistance to Standard therapy more than 2 months
5. Informed consent

Exclusion Criteria:

1. Congenital Heart Disease
2. Active infection less than one month
3. Dysrhythmia
4. Cardiogenic shock
5. Renal failure
6. Immune Deficiency (Documentation)
7. Terminal illness or malignancy(Documentation)
8. TORCH (Documentation)
9. Metabolic disorder (Documentation)
10. Neuromuscular disorder (Documentation)
11. Autoimmune disease (Documentation)
12. Developmental delay
13. Cytotoxic drugs
14. Previous bone marrow transplant
15. Contraindications to CMR such as metallic implants

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Death | 3months
  The rate of patients' death 3 months after cell transplantation
Arrest | 3 months
  The rate of patients' arrests 3 months after cell transplantation

SECONDARY OUTCOMES:
Dysrhythmia | 3 months
  The rate of dysarthymia 3 months after cell transplantation
Heart transplantation | 3 months
  The rate of demand for heart transplantation 3 months after cell transplantation.
Hospital admission for heart failure | 3 months
  The rate of hospital administration 3 months after cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine & Cell therapy center of Royan Institute; Mohammad Mahdavi, MD, Study Director — Department of Pediatric Cardiology, Rajaie Cardiovascular Medical and Research Center, Iran University of Medical Sciences, Tehran, Iran; Koorosh Vahidshahi, MD, Principal Investigator — Department of Pediatric Cardiology, Rajaie Cardiovascular Medical and Research Center, Iran University of Medical Sciences, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org